CLINICAL TRIAL: NCT05742334
Title: RAP: Prospective Pilot Trial Evaluating Return to Continence and Potency Following Radical Prostatectomy Using Novel Multi-Layer Perinatal Tissue Allograft
Brief Title: Evaluating Return to Continence and Potency Following Radical Prostatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor decided to not move forward with this study
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Samaritan Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00093386; WFBCCC 85321 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2023-02-02; First posted 2023-02-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Bladder continence after prostatectomy; Erectile function after prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Robot Assisted Radical Prostatectomy with MLG-COMPLETE Allograft (Experimental): Implantation of the MLG-COMPLETE allograft during your robot-assisted radical prostatectomy surgery.
  Interventions: Procedure: Robot-Assisted Radical Prostatectomy with MLG-COMPLETE Allograft Implantation; Device: MLG-COMPLETE Allograft Implantation

INTERVENTIONS:
Procedure: Robot-Assisted Radical Prostatectomy with MLG-COMPLETE Allograft Implantation — The intervention will be administered on an inpatient basis. Participants receiving MLG-Complete™ will have it placed around the neurovascular bundle. Placement of the graft should not take more than 5 minutes, therefore, there should be minimal impact to overall surgical time.
Device: MLG-COMPLETE Allograft Implantation — The MLG-Complete™ allograft will be placed on each neurovascular bundle (NVB) bilaterally as shown on the above picture after excision of the prostate prior to completing the urethrovesical anastomosis.

SUMMARY:
The purpose of this research is to determine if using human placental membrane (also called an allograft) helps to improve recovery time for erectile function and bladder control after having robot-assisted radical prostatectomy (RARP) surgery.

DETAILED DESCRIPTION:
Primary Objective(s):

* To evaluate the safety and feasibility of MLG-Complete™ allograft placement in patients who undergo robot-assisted radical prostatectomy (RARP) with bilateral nerve sparing.
* To determine the effectiveness of using MLG-Complete™ allograft to optimize return to erectile function (potency) in patients who have had robot-assisted radical prostatectomy (RARP) with bilateral nerve sparing by utilizing the Sexual Health Inventory for Men (SHIM) score.
* To determine the effectiveness of using MLG-Complete™ allograft to optimize return to continence in patients who have had robot-assisted radical prostatectomy (RARP) with bilateral nerve sparing by utilizing the American Urological Association (AUA) symptom score, assessing daily pad use from direct patient report, and by utilizing the International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI Short Form).

OUTLINE: Patients undergo RARP with placement of the MLG-Complete allograft on study.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects age 40 to 70.
* Primary diagnosis of untreated clinically localized prostate cancer as defined by histopathological diagnosis by prostate biopsy and cross sectional imaging, as indicated based on guidelines.
* Planned elective robot-assisted radical prostatectomy with bilateral nerve sparing technique for clinically localized prostate cancer.
* Urine bacterial culture should be negative for infection within 30 days of surgery.
* Patient has no erectile dysfunction (Sexual Health Inventory for Men [SHIM] Score >17) prior to the date of surgery.
* Patient is willing to follow study procedures and complete follow-up surveys.
* Patient has the ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Patients with high-risk prostate cancer planned for neoadjuvant therapy, full or partial excision of neurovascular bundles.
* Patient is unable to document penile rehabilitation, including oral 5-phosphodiesterase inhibitor use, vacuum pump therapy use, and/or injectable medications.
* Patients who received treatment with immuno-suppressants (including systemic corticosteroids) within two weeks prior to surgery or those who anticipate requiring immunosuppressive treatment during the study.
* Patients who received cytotoxic chemotherapy within one month prior to initial screening, or who receive this treatment during the screening period, or who are anticipated to require treatment during the course of the study.
* Patients that have had prior hormonal therapy such as Lupron or oral anti-androgens.
* Patients with poor urinary control at baseline requiring the use of pads for leakage.
* Previous history of pelvic radiation.
* Previous history of simple prostatectomy or transurethral prostate surgery.
* Patients with obesity defined as body mass index > 40 kg/m2.
* History of open pelvic surgery except for hernia repair.
* Patients with diabetes.
* Patients scheduled at the time of screening to undergo chemotherapy, radiation, hormone therapy, or open surgery during the study period.
* Neurologic or psychiatric disorders that may confound postsurgical assessments determined at the discretion of the investigator.
* Received administration of an investigational drug within 30 days prior to study, and/or has planned administration of another investigational product or procedure during participation in this study.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events Using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to 12 months
  Safety will be assessed by describing the frequency and nature of adverse events using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 throughout the study
Number of Adverse Events Using the Clavien-Dindo Classification System | Up to 12 months
  Adverse effects per the Clavien-Dindo Classification system will be assessed descriptively post-graft placement The Clavien-Dindo system is widely used throughout surgery for grading adverse events (i.e. complications) which occur as a result of surgical procedures. It consists of 7 grades.
  Grade I - Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions; Grade II - Requiring pharmacological treatment with drugs other than such allowed for grade I complications Grade III - Requiring surgical, endoscopic or radiological intervention
  * IIIa - Intervention not under general anesthesia
  * IIIb - Intervention under general anesthesia; Grade IV - Life-threatening complication (including central nervous system complications) requiring intensive care/intensive care unit-management
  * IVa - single organ dysfunction (including dialysis)
  * IVb - Multi-organ dysfunction and Grade V - Death
Number of Participants Screened for Enrollment | Up to 12 months
  Feasibility will be assessed by determining the number of patients screened in order to enroll the anticipated number of participants to study intervention.
Number of Participants to Complete Intervention | Up to 12 months
  Rates of completion will be determined at each visit based on the anticipated number of participants to study intervention that complete each visit.
Average Time for Participants to Return to Potency - Sexual Health Inventory for Men (SHIM) Questionnaire | Up to 12 months
  Return to potency will be defined as the time to attain the ability to achieve an erection sufficient for intercourse >50% of the time or at least 50% rigidity compared to baseline status post robot-assisted radical prostatectomy using the Sexual Health Inventory for Men (SHIM) questionnaire. This questionnaire is used to diagnose erectile dysfunction (ED) and severity as moderate score ranging 8-11, mild to moderate 12-16, 17-21 mild, and 22-25 no ED
Average Time to Return to Bladder Control/Urinary Continence - ICIQ-UI Short Form | Up to 12 months
  effectiveness will be measured by the average time for return to continence as defined as the time from radical prostatectomy to until the use of < 1 incontinence pad and by the and by the ICIQ-UI Short Form. This tool is a four-item questionnaire to objectively evaluate urinary incontinence (UI) and its associated impact on quality of life. Scores range from 0-21 with a higher score indicating greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok K Hemal, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No